CLINICAL TRIAL: NCT04633512
Title: Safety and Feasibility of ActivSightTM Laser Speckle Imaging in Visualization of Tissue Perfusion and Vasculature in Human
Brief Title: Safety and Feasibility of ActivSightTM in Human
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Activ Surgical (Industry)
Collaborators: The University of Texas Health Science Center, Houston (Other); University at Buffalo (Other); Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ACF0012020
Record Dates: First submitted 2020-10-28; First posted 2020-11-18 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Acute Cholecystitis; Colorectal Cancer; Diverticulitis, Colonic; Obesity, Morbid; Inflammatory Bowel Diseases
Keywords: laparoscopic; robot assisted surgery; gastrointestinal anastomoses; cholecystectomy; colorectal surgery; bariatric surgery; vascularity; perfusion; ICG; laser speckle contrast imaging
MeSH Terms: conditions — Cholecystitis, Acute; Colorectal Neoplasms; Diverticulitis, Colonic; Obesity, Morbid; Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: Target enrollment is 80 patients. Feasibility will be studied under two categories of operations: feasibility in patients undergoing intestinal anastomoses for bariatric or colorectal surgery (n=52); and feasibility in patients undergoing cholecystectomy (n=28).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- ActivSight Group (Experimental): Patients undergoing intestinal anastomoses (colorectal and bariatric) with ActivSight (n=52) Patients undergoing cholecystectomy with ActivSight (n=28)
  Interventions: Device: ActivSight

INTERVENTIONS:
Device: ActivSight — Use of ActivSight in patients undergoing laparoscopic or robot assisted intestinal anastomoses and patients undergoing laparoscopic or robot assisted cholecystectomy.

SUMMARY:
ActivSightTM combines an innovative form factor and proprietary software to deliver precise, objective, real-time visualization of blood flow and tissue perfusion intraoperatively for laparoscope-based surgery. A small adaptor that fits between any existing laparoscope and camera systems and a separate light source placed along any current commercial system will deliver objective real-time tissue perfusion and blood flow information intraoperatively.

Primary Objective: To determine safety and feasibility of ActivSightTM in displaying tissue perfusion in intestinal anastomoses including colorectal and bariatric surgery.

Secondary Objective: To determine the efficacy of ActivSightTM in; (1) displaying tissue vascularity and perfusion in comparison to indocyanine green (ICG) during gastrointestinal anastomoses; and (2) displaying biliary tree during laparoscopic cholecystectomy using ICG-based intraoperative cholangiography (IOC).

DETAILED DESCRIPTION:
Design:

* This is a feasibility study designed to evaluate safety and feasibility of ActivSightTM in gastrointestinal anastomoses and cholecystectomy.
* Safety will be determined through clinical assessments and evaluation of any adverse event.
* Feasibility will be determined through technically successful completion of intended visualization.
* Assessment of preliminary efficacy will be performed through analysis of any intraoperative decisions made based on visual display as compared to standard endoscopic approach, or non-inferiority to ICG-based visualization and usability.
* Patients outcome and follow up to Postoperative day 28 will be monitored for clinical outcome.
* Target enrollment for the assessment of 80 patients; 52 evaluating intestinal anastomoses cases (including bariatric and colorectal cases); and 28 evaluating laparoscopic cholecystectomy. Stopping rules are triggered following the first 6 patients and a comparison group 6 patients in ICG-based treatment.

ELIGIBILITY:
Inclusion Criteria:

* All patients age >= 18 years old undergoing laparoscopic or robot assisted intestinal anastomoses, or all patients age >= 18 years old who are planned for laparoscopic cholecystectomy; spoken command and literacy in the native language spoken at each participating center; ability to understand and follow study procedures; and having provided signed consent.
* Diagnosis:
* All patients with a clinical suspicion and diagnosis of benign or malignant, small or large bowel lesions requiring surgical resection.
* All patients with clinical suspicion and diagnosis of symptomatic cholelithiasis or cholecystitis planned for cholecystectomy.
* Typical imaging as per standard workup findings including US, CT and/or MRI. Plain radiographs and contrast imaging may be obtained by referring physicians and are helpful for confirming the clinical diagnosis.
* Any bariatric patients undergoing gastric sleeve or bypass.
* Any pediatric patient undergoing laparotomy for necrotizing enterocolitis
* Location of pathology or resected segment:
* Target lesions can be located in any fore-, mid- or hindgut segments requiring reconstruction and anastomoses.
* Prior therapy:
* Patients with prior surgery are eligible for enrollment.
* Laboratory:
* Hemoglobin > 9 g/dL
* Platelet count ≥75,000/μL (may receive transfusions)
* Normal prothrombin time, tested prothrombin, and international normalized ratio < 1.5 x upper limit of normal (ULN) (including patients on prophylactic anticoagulation)
* Renal function: Age-adjusted normal serum creatinine derived from Schwartz formula for estimating glomerular filtration rate by the Centers for Disease Control (CDC) or a creatinine clearance ≥60 mL/min/1.73 m2 for safe
* Adequate pulmonary function: Defined as no dyspnea at rest, and a pulse oximetry >94% on room air if there is clinical indication for determination.

Exclusion Criteria:

* There is no exclusion criteria for ActivSightTM for gastrointestinal resection.
* Patients assigned to FDA cleared ICG-based visualization are contraindicated for any chronic renal dysfunction, potential drug interaction, history of allergy to ICG or anaphylaxis, and pregnancy.
* Patients eligible for cholecystectomy, exclusion criteria include known allergy to iodides; known history of cholangitis, pancreatitis, prior common bile duct injury, coagulopathy or known, preexisting liver disease; pregnancy or breast-feeding; or being of reproductive age with pregnancy possible and not ruled out.
* Patients currently in any investigational agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2020-11-17 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events in 28 days following use of ActivSightTM | 28 days
  To determine safety of ActivSightTM in patients undergoing intestinal anastomoses, as defined through clinical assessments and evaluation of use related adverse events intraoperatively and a routine follow up at 28 days following surgery. ActivSightTM will be deemed safe if hardware (adaptor or light source)-related major (serious) adverse event is encountered in the treated patients and if less than 2 hardware-related minor adverse events are encountered.
  Adverse events will be summarized descriptively and tabulations on the type, severity, and relationship to application will be performed and any changes of outcomes from baseline on follow up will be examined using the nonparametric Wilcoxon rank test.
Preparation time of ActivSightTM. | 1 day
  Rate on a scale of 1-5 (1 = Difficult to use or Unsatisfied - 5 = no training required or very satisfied): How easy was ActivSight to set up?
Latency of display of ActivSightTM. | 1 day
  Rate on a scale of 1-5 (1 = Difficult to use or Unsatisfied - 5 = no training required or very satisfied): How specifically did ActivSight display the intended field and the target tissue of interest?
Resolution of display of ActivSightTM. | 1 day
  Rate on a scale of 1-5 (1 = Difficult to use or Unsatisfied - 5 = no training required or very satisfied): How was the display quality of ActivSight on the intended field and target tissue of interest?
Specificity of display of ActivSightTM. | 1 day
  Specificity of display will serve as an outcome for feasibility. Yes/No question for surgeon: "Does the perfusion information displayed by ActivSightTM reflect the expected pattern of blood flow interruption?"
Usability of ActivSightTM by surgeon, as quantified by Likert scale. | 1 day
  Likert scale ratings will serve as an outcome for feasibility. Scale 1-5 question (1=strongly disagree, 2=slightly disagree, 3=neutral, 4=slightly agree, 5=strongly agree): "ActivSightTM was easy to use while operating."
Support personnel satisfaction with ActivSightTM, as quantified by Likert scale. | 1 day
  Likert scale ratings will serve as an outcome for feasibility. Scale 1-5 question (1=strongly disagree, 2=slightly disagree, 3=neutral, 4=slightly agree, 5=strongly agree): "ActivSightTM was easy to set up for the procedure."

SECONDARY OUTCOMES:
Ability of ActivSightTM to display perfusion. | 1 day
  ActivSightTM ability to display perfusion at a tissue level during gastrointestinal anastomoses is measured by the following Yes/No question for the surgeon: "Does ActivSightTM display tissue perfusion of the anatomy during anastomoses in comparison to ICG?"
Ability of ActivSightTM to display blood vessels. | 1 day
  ActivSightTM ability to display blood vessels during gastrointestinal anastomoses is measured by the following Yes/No question for the surgeon: "Does ActivSightTM display vascularity of the anatomy during anastomoses in comparison to ICG?"
Ability of ActivSightTM to display biliary tree. | 1 day
  The clinical metrics for displaying biliary tree will be evaluated using the following question: "Which of the following biliary structures are you able to identify using ActivSightTM with ICG? (Select all that apply): common bile duct (CD), right hepatic duct (RHD), common hepatic duct (CHD), common bile duct (CBD), cystic common bile duct junction (CCBDJ), cystic gallbladder junction (CGJ), accessory ducts (AD)."

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Kaleida Health, University of Buffalo, Buffalo, New York
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Memorial Hermann Sugar Land Hospital, Sugar Land, Texas

DOCUMENTS (1):
  • Study Protocol (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/12/NCT04633512/Prot_000.pdf